CLINICAL TRIAL: NCT07103707
Title: Comparison of Frequency of Wound Infection Between Open and Laparoscopic Cholecystectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Reading Hospital, Pakistan (Other Government)
Responsible Party: Principal Investigator, Moeez u din Khan, surgical resident, Lady Reading Hospital, Pakistan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 253/LRH/MTI
Record Dates: First submitted 2025-07-11; First posted 2025-08-05 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-08

CONDITIONS: Wound Infection, Surgical
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Intervention Model Description: randomization will performed by blocked randomization (61 in each group) 61 patient will be in open cholecystectomy group( A )while 61 patient will be in laparoscopic cholecystectomy group (B)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- open cholecystectomy (Active Comparator): patient undergoing open cholecystectomy
  Interventions: Procedure: open cholecystectomy
- laparoscopic cholecystectomy (Active Comparator): patient undergoing laparoscopic cholecystectomy
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: open cholecystectomy — standard open cholecystectomy performed under general anesthesia
  Arms: open cholecystectomy
Procedure: Laparoscopic cholecystectomy — Standard laparoscopic cholecystectomy using minimally invasive technique
  Arms: laparoscopic cholecystectomy

SUMMARY:
The goal of this clinical trial is to compare the frequency of wound infection between open and laparoscopic cholecystectomy in adult patient aged 18- 65 years with symptomatic cholelithiasis admitted through OPD the main question it aims to answer are

* Does there is difference in the frequency of wound infection in patients with open cholecystectomy as compared to laparoscopic cholecystectomy Researcher will compare the frequency of wound infection in participant undergoing open and laparoscopic cholecystectomy to see there is difference in frequency of wound infection between open and laparoscopic cholecystectomy Participants will be asked
* To Visit OPD after 1 week for follow up
* Keep record of symptoms like erythema, pain, cloudy drainage from the incision site

ELIGIBILITY:
Inclusion Criteria:

* Both genders

  * Patients aged 18 to 65 years
  * Symptomatic cholelithiasis as per operational definition
  * Undergoing cholecystectomy (open/laparoscopic)
  * ASA score I/II (Annexure-II)

Exclusion Criteria:

* ● H/o diabetes mellitus

  * H/o immunocompromised state (e.g. HIV, steroid use)
  * H/o acute cholecystitis
  * H/o empyema gallbladder
  * H/o gallbladder perforation ● H/o choledocholithiasis
  * H/o portal hypertension
  * H/o abnormal blood clotting profiles (PTT >15 seconds, APTT >20 seconds)
  * H/o pregnancy on HCG

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
comparison of frequency of wound infection between open and laparoscopic cholecystectomy | 1 year
  to compare the frequency of wound infection in patients undergoing open and laparoscopic

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad faraz, AP GS(FCPS), Principal Investigator — Lady reading hospital peshawar
Locations (1):
- Moeez u din khan, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: No